CLINICAL TRIAL: NCT02225834
Title: Effects of Early Atorvastatin Treatment During the Acute Phase of Stroke on Immunoinflammatory Markers and Outcome in Patients With Acute Ischemic Stroke Classified as LAAS According TOAST Classification
Brief Title: Atorvastatin in Acute Stroke Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Antonino Tuttolomondo, Assistant Professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21770
Record Dates: First submitted 2014-03-11; First posted 2014-08-26 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Ischemic Stroke
Keywords: Atorvastatin, ischemic stroke, cytokines
MeSH Terms: conditions — Ischemic Stroke | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- early Atorvastatin treatment (Experimental): Ischemic stroke patients treated with with atorvastatin 80 mg at admission until discharge
  Interventions: Drug: Atorvastatin
- no early treatment with atorvastatin (No Intervention): Ischemic stroke patients not treated with with atorvastatin 80 mg until discharge

INTERVENTIONS:
Drug: Atorvastatin — treatment with atorvastatin 80 mg (once-daily) from admission day until discharge
  Arms: early Atorvastatin treatment

SUMMARY:
Recent clinical trials and meta-analyses of b-hydroxy-bmethylglutaryl coenzyme A (HMG-CoA) reductase inhibitors (statins) have demonstrated a significant reduction in ischemic stroke in patients with a history of coronary artery disease, both with and without elevations of serum cholesterol. Recent data suggest that statins have other beneficial properties in addition to the retardation of atherosclerosis. Asahi et al demonstred that Statins increased eNOS and tPA mRNA levels but did not change mRNA levels of PAI-1 and that In eNOS knockout mice, atorvastatin reduced the volume of ischemic tissue and improved neurologic outcomes after arterial occlusion by blood clot emboli. In addition to their lipid-lowering effects, it has been speculated that statins may also have beneficial effects on cerebral circulation and brain parenchyma during ischaemic stroke and reperfusion. Aslanyan et al reported that statin use was associated with reduced mortality at 1 month during the follow-up.

In patients with recent stroke or TIA and without known coronary heart disease, 80 mg of atorvastatin per day reduced the overall incidence of strokes and of cardiovascular events, despite a small increase in the incidence of hemorrhagic stroke period .

Recently the investigators group reported that lacunar strokes compared to nonlacunar ones exhibited significantly lower plasma levels of TNF-α and IL1-β, P-selectin and ICAM-1 24-72 h and 7-10 days after stroke onset (4). At extracranial arterial territories, inflammation plays a crucial role mediating all the stages of the atherosclerosis process . Similarly, thrombosis and defective fibrinolysis may also contribute to the progression of atherosclerotic lesions . Interestingly, both mechanisms might have a relevant role in the pathogenesis of intracranial large artery atherosclerosis and ischemic stroke Moreover our group showed that Patients with cardioembolic and atherothrombotic stroke subtypes showed significantly higher median plasma levels of TNF-α, IL-6, IL-1β whereas the lacunar subtype showed significantly lower median plasma levels of TNF-α, IL-6 and IL-1β and that immunoinflammatory marker plasma levels are significantly related to ischemic lesion volume.

A meta-analysis showed that statins may possess antithrombotic property because these drugs were reported to reduce periprocedural infarction in patients undergoing percutaneous coronary intervention .

This clinical benefit was detected after median, 0.5 days of treatment with statins (indicating that statins could potentially exert an antithrombotic effect even earlier than supposed from pharmacological studies.

Violi et al recently showed the first evidence that atorvastatin acutely and simultaneously decreases oxidative stress and platelet activation by directly inhibiting platelet Nox2 and ultimately platelet isoprostanes and thromboxane A2 so providinf a rationale for the use of statins to prevent or modulate coronary thrombosis.

Whereas recent data suggest that inflammatory reactions are involved in the pathogenesis and progression of cerebral ischaemia , no study has evaluated effects of atorvastatin 80 mg/day after a recent stroke on stroke outcome and on immunoinflammatory markers so to evaluate acute antithrombotic and anti-inflammatory effects of atorvastatin also in acute cerebrovascular event setting.

On this basis the primary objective of the study was to evaluate the separate effects of atorvastatin in vivo on immunoinflammatory markers and on stroke prognosis in patients with recent acute ischemic stroke classified as atherothrombotic.

DETAILED DESCRIPTION:
Material and Methods The investigators will enroll patients with a diagnosis of acute ischemic stroke admitted to the Internal Medicine Department at the University of Palermo between November 2011 and October 2014. The controlsubjects were patients admitted, in the same period, to our Internal Medicine Department for any cause different from acute cardiovascular and cerebrovascular events or exclusion criteria. Every subject with ischemic stroke was matched for age (±3 years), sex, and cardiovascular risk factor prevalence with one control subject

Study Hypothesis and Patient Population:

The primary hypothesis of the study is that treatment with 80 mg of atorvastatin per day administered early at admission after acute ischemic stroke would reduce immunoinflammatory activation of the acute phase and that this immunoinflammatory modulation could have a possible effect on prognosis of ischemic stroke evaluated by some outcome indicators.

Eligible patients are men and women over 18 years of age who had an acute ischemic stroke Patients with inflammatory or infectious diseases, cancer, hematological diseases and severe renal or liver failure, as well as those who were under treatment with anti-inflammatory will be excluded Stroke was defined by focal neurological signs or symptoms thought to be of vascular origin that persisted for >24 h, confirmed by brain CT and/or MRI in baseline conditions Cardiovascular risk factors will be evaluated for both subjects and controls on the basis of the following criteria: type 2 diabetes will be determined using a clinically based algorithm that considered age at onset, presenting weight and symptoms, family history, onset ofinsulin treatment, and history of ketoacidosis. Atrial fibrillation will be diagnosed when present on the admission ECG. Hypertension was present when a patient had received antihypertensive treatment before admission or when hypertension was diagnosed during the hospital stay by repeated detection of blood pressure ≥160/95 mmHg. Hypercholesterolemia was defined as total serum cholesterol ≥200 mg/dl or on the basis of a clinical history of hypercholesterolemia or statin treatment.

The studyIs pending of approvationby the Ethics Committee of the "Policlinico P. Giaccone" of Palermo. Written informed consent wasobtained for all patients.

The type of acute ischemic stroke will be classified according to the TOAST classification (Adams et al., 1993): 1) Large Artery Athero- Sclerosis (LAAS); 2) CardioEmbolic Infarct (CEI); 3) LACunar infarct (LAC); 4) stroke of Other Determined Etiology (ODE); 5) stroke of UnDetermined Etiology (UDE).

• Large artery atherosclerosis (LAAS) These patients will have clinical and brain imaging findings of either significant (≥50%) stenosis or occlusion of a major brain artery or branch cortical artery, presumably due to atherosclerosis. Clinical findings include those of cerebral cortical impairment (aphasia, neglect, restricted motor involvement, etc.) or brain stem or cerebellar dysfunction. Cortical or cerebellar lesions and brain stem or subcortical hemispheric infarcts greater than 1.5 cm in diameter on CT or MRI are considered to be of potential large artery atherosclerotic origin. Supportive evidence by duplex imaging or arteriography of a stenosis of greater than 50% of an appropriate intracranial or extracranial artery is needed. Diagnostic studies should exclude potential sources of cardiogenic embolism.

Patient evaluation and blood sample collection All the ischemic stroke patients will undergo: medical history with recordi ng of potential stroke risk factors, blood and coagulation tests, 12-lead ECG, 24 h electrocardiography monitoring, trans-thoracic echocardiography, carotid ultrasound, brain CT or MRI at admission (repeated between the third and the seventh days of stroke onset).

Blood samples will be obtained in the non-fasting state. After 10 min of rest in the supine position, vital signs were recorded and blood samples were collected from the antecubital vein. EDTA-anticoagulated peripheral blood was drawn from each patient within 12 h from symptom onset. Serum and plasma were immediately separated by centrifugation and stored in aliquots at -80 °C until analysis.

The investigators will evaluate plasma levels of IL-1β, TNF-α, IL-6 and IL-10, Eselectin, P-selectin, sICAM-1 and sVCAM-1 as markers of immunoinflammatory activation, VWF plasma levels as a marker of endothelial dysfunction, TPA-antigen and PAI-1 plasma levels as thrombotic/ fibrinolytic markers.

These laboratory evaluation will be done at 72 h and at one week after symptom onset.

IL-1β, TNF-α, IL-6 and IL-10 and VWFantigen were measured using a sandwich ELISA (Human IL-1β, TNF-α, IL-6 and IL-10 Quantikine, R&D Systems (VWF ELISA kitdurian, Instrumentation Laboratory, Milano, Italy); VCAM-1, ICAM-1, E-selectin, P-selectin, PAI-1 and TPAantigen will be measured by commercial bioimmunoassay (Human sICAM-1, sVCAM-I, sE-selectin and sP-selectin Parameter, Quantikine, R&D Systems, Gentaur AssayMax Human Plasminogen Activator Inhibitor-1 (PAI-1) ELISA Kit, Gentaur AssayMax Tissue Plasminogen Activator (TPA) ELISA Kit).

The minimum detectable concentrations for the diagnostic tests were: TNF alpha: 1.6 pg/mL, IL-1β: b1 pg/mL; IL-6:b0.70 pg/mL; IL-10: N3.9 pg/mL; ICAM-1:b0.35 ng/mL;VCAM-1:0.6 ng/mL; E-Selectin: b0.1 ng /mL; P-Selectin:b0.5 ng/mL; vWF:1.0%;TPA: 0.3 pg/ml; PAI-1: b50 pg/ml. Intra-assay and inter-assay coefficients of variation were: TNF alpha: 4.2% and 4.6%; IL-1β: 3.3% and 4.2%; IL-6: 1.6% and 3.3%; IL-10: 4.3% and 7.5%; ICAM-1: 4.8% and 6.1%; VCAM-1: 3.5% and 7.7%; ESelectin: 4.8% and 5.7%; P-Selectin: 4.9% and 8.8%; vWF: 5% and 10%; TPA: 4.8% and 5%; PAI-1: 5.7% and 8.3%.

As outcome indicators the investigators will use evaluation of acute neurological deficit by means National Institutes of Health Stroke Scale, at 72 hours and 7 days after admission and evaluation of disability at 7 days after admission by means modified Rankin Scale Neurological deficit score on admission was evaluated by the NIHSS. The National Institutes of Health Stroke Scale, or NIH Stroke Scale (NIHSS) is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0 Disability at 7 days was evaluated by modified Rankin Scale (mRS) that is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke.

The scale runs from 0-6, running from perfect health without symptoms to death.

* 0 - No symptoms.
* 1 - No significant disability. Able to carry out all usual activities, despite some symptoms.
* 2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
* 3 - Moderate disability. Requires some help, but able to walk unassisted.
* 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
* 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
* 6 - Dead. Treatment protocol

Patients will be randomized to these two treatment:

Group A: treatment with atorvastatin 80 mg (once-daily) from admission day until discharge Group B: No treatment with atorvastatin 80 mg until discharge, after discharge treatment with atorvastatin 80 mg will be started

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were men and women over 18 years of age who had an acute ischemic stroke with a symptom time onset < 48 hours

Exclusion Criteria:

* Patients with inflammatory or infectious diseases, cancer, hematological diseases and severe renal or liver failure, as well as those who were under treatment with anti-inflammatory were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-11; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
NIHSS score at 72 hour | 72 hours
  differences with regard of NIHSS score at 72 hours
differences in msRankin score | 72 hours

SECONDARY OUTCOMES:
Plasma levels of inflammatory cytokines at 72 hours | 72 hours
  differences with regard of plasma levels of TNF-alfa, IL-1 beta, IL-6, E-Selectin, P-Selectin, ICAM-1, V-CAM1, VWF
Outcome measure ( rankin score) | seven days
  differences in msRankin score at seven day after admission

CONTACTS AND LOCATIONS:
Locations (1):
- Internal Medicine Ward, University of Palermo, Palermo, Italy, Italy

REFERENCES:
- [Background] Asahi M, Huang Z, Thomas S, Yoshimura S, Sumii T, Mori T, Qiu J, Amin-Hanjani S, Huang PL, Liao JK, Lo EH, Moskowitz MA. Protective effects of statins involving both eNOS and tPA in focal cerebral ischemia. J Cereb Blood Flow Metab. 2005 Jun;25(6):722-9. doi: 10.1038/sj.jcbfm.9600070. PMID 15716855
- [Background] Aslanyan S, Weir CJ, McInnes GT, Reid JL, Walters MR, Lees KR. Statin administration prior to ischaemic stroke onset and survival: exploratory evidence from matched treatment-control study. Eur J Neurol. 2005 Jul;12(7):493-8. doi: 10.1111/j.1468-1331.2005.01049.x. PMID 15958087
- [Background] Amarenco P, Bogousslavsky J, Callahan A 3rd, Goldstein LB, Hennerici M, Rudolph AE, Sillesen H, Simunovic L, Szarek M, Welch KM, Zivin JA; Stroke Prevention by Aggressive Reduction in Cholesterol Levels (SPARCL) Investigators. High-dose atorvastatin after stroke or transient ischemic attack. N Engl J Med. 2006 Aug 10;355(6):549-59. doi: 10.1056/NEJMoa061894. PMID 16899775
- [Background] Licata G, Tuttolomondo A, Corrao S, Di Raimondo D, Fernandez P, Caruso C, Avellone G, Pinto A. Immunoinflammatory activation during the acute phase of lacunar and non-lacunar ischemic stroke: association with time of onset and diabetic state. Int J Immunopathol Pharmacol. 2006 Jul-Sep;19(3):639-46. doi: 10.1177/039463200601900320. PMID 17026849
- [Background] Tuttolomondo A, Di Sciacca R, Di Raimondo D, Serio A, D'Aguanno G, La Placa S, Pecoraro R, Arnao V, Marino L, Monaco S, Natale E, Licata G, Pinto A. Plasma levels of inflammatory and thrombotic/fibrinolytic markers in acute ischemic strokes: relationship with TOAST subtype, outcome and infarct site. J Neuroimmunol. 2009 Oct 30;215(1-2):84-9. doi: 10.1016/j.jneuroim.2009.06.019. Epub 2009 Aug 19. PMID 19695716
- [Background] Licata G, Tuttolomondo A, Di Raimondo D, Corrao S, Di Sciacca R, Pinto A. Immuno-inflammatory activation in acute cardio-embolic strokes in comparison with other subtypes of ischaemic stroke. Thromb Haemost. 2009 May;101(5):929-37. PMID 19404547
- [Background] Pignatelli P, Carnevale R, Pastori D, Cangemi R, Napoleone L, Bartimoccia S, Nocella C, Basili S, Violi F. Immediate antioxidant and antiplatelet effect of atorvastatin via inhibition of Nox2. Circulation. 2012 Jul 3;126(1):92-103. doi: 10.1161/CIRCULATIONAHA.112.095554. Epub 2012 May 21. PMID 22615342
- [Background] Iadecola C, Anrather J. The immunology of stroke: from mechanisms to translation. Nat Med. 2011 Jul 7;17(7):796-808. doi: 10.1038/nm.2399. PMID 21738161
- [Background] Yilmaz G, Granger DN. Leukocyte recruitment and ischemic brain injury. Neuromolecular Med. 2010 Jun;12(2):193-204. doi: 10.1007/s12017-009-8074-1. Epub 2009 Jul 5. PMID 19579016
- [Background] Konsman JP, Drukarch B, Van Dam AM. (Peri)vascular production and action of pro-inflammatory cytokines in brain pathology. Clin Sci (Lond). 2007 Jan;112(1):1-25. doi: 10.1042/CS20060043. PMID 17132137
- [Background] Sairanen TR, Lindsberg PJ, Brenner M, Siren AL. Global forebrain ischemia results in differential cellular expression of interleukin-1beta (IL-1beta) and its receptor at mRNA and protein level. J Cereb Blood Flow Metab. 1997 Oct;17(10):1107-20. doi: 10.1097/00004647-199710000-00013. PMID 9346436
- [Background] Blum A, Shamburek R. The pleiotropic effects of statins on endothelial function, vascular inflammation, immunomodulation and thrombogenesis. Atherosclerosis. 2009 Apr;203(2):325-30. doi: 10.1016/j.atherosclerosis.2008.08.022. Epub 2008 Sep 2. PMID 18834985
- [Background] Antoniades C, Bakogiannis C, Leeson P, Guzik TJ, Zhang MH, Tousoulis D, Antonopoulos AS, Demosthenous M, Marinou K, Hale A, Paschalis A, Psarros C, Triantafyllou C, Bendall J, Casadei B, Stefanadis C, Channon KM. Rapid, direct effects of statin treatment on arterial redox state and nitric oxide bioavailability in human atherosclerosis via tetrahydrobiopterin-mediated endothelial nitric oxide synthase coupling. Circulation. 2011 Jul 19;124(3):335-45. doi: 10.1161/CIRCULATIONAHA.110.985150. Epub 2011 Jul 5. PMID 21730307
- [Background] Santos MT, Fuset MP, Ruano M, Moscardo A, Valles J. Effect of atorvastatin on platelet thromboxane A(2) synthesis in aspirin-treated patients with acute myocardial infarction. Am J Cardiol. 2009 Dec 15;104(12):1618-23. doi: 10.1016/j.amjcard.2009.07.039. PMID 19962464
- [Background] Pignatelli P, Sanguigni V, Lenti L, Loffredo L, Carnevale R, Sorge R, Violi F. Oxidative stress-mediated platelet CD40 ligand upregulation in patients with hypercholesterolemia: effect of atorvastatin. J Thromb Haemost. 2007 Jun;5(6):1170-8. doi: 10.1111/j.1538-7836.2007.02533.x. PMID 17388962
- [Background] Nakamura K, Masuda H, Kariyazono H, Arima J, Iguro Y, Yamada K, Sakata R. Effects of atorvastatin and aspirin combined therapy on inflammatory responses in patients undergoing coronary artery bypass grafting. Cytokine. 2006 Dec;36(5-6):201-10. doi: 10.1016/j.cyto.2006.11.001. Epub 2007 Feb 14. PMID 17300951
- [Background] Moonis M, Kane K, Schwiderski U, Sandage BW, Fisher M. HMG-CoA reductase inhibitors improve acute ischemic stroke outcome. Stroke. 2005 Jun;36(6):1298-300. doi: 10.1161/01.STR.0000165920.67784.58. Epub 2005 May 5. PMID 15879346
- [Background] Reis PA, Estato V, da Silva TI, d'Avila JC, Siqueira LD, Assis EF, Bozza PT, Bozza FA, Tibirica EV, Zimmerman GA, Castro-Faria-Neto HC. Statins decrease neuroinflammation and prevent cognitive impairment after cerebral malaria. PLoS Pathog. 2012 Dec;8(12):e1003099. doi: 10.1371/journal.ppat.1003099. Epub 2012 Dec 27. PMID 23300448
- [Background] Piermartiri TC, Figueiredo CP, Rial D, Duarte FS, Bezerra SC, Mancini G, de Bem AF, Prediger RD, Tasca CI. Atorvastatin prevents hippocampal cell death, neuroinflammation and oxidative stress following amyloid-beta(1-40) administration in mice: evidence for dissociation between cognitive deficits and neuronal damage. Exp Neurol. 2010 Dec;226(2):274-84. doi: 10.1016/j.expneurol.2010.08.030. Epub 2010 Sep 15. PMID 20816828
- [Derived] Tuttolomondo A, Di Raimondo D, Pecoraro R, Maida C, Arnao V, Della Corte V, Simonetta I, Corpora F, Di Bona D, Maugeri R, Iacopino DG, Pinto A. Early High-dosage Atorvastatin Treatment Improved Serum Immune-inflammatory Markers and Functional Outcome in Acute Ischemic Strokes Classified as Large Artery Atherosclerotic Stroke: A Randomized Trial. Medicine (Baltimore). 2016 Mar;95(13):e3186. doi: 10.1097/MD.0000000000003186. PMID 27043681